CLINICAL TRIAL: NCT06032572
Title: Evaluation of the Safety and Effectiveness of the VRS100 Robotic Console System in Percutaneous Coronary Interventions: A Multicenter, Randomised, Non-inferiority Trial (ESSENCE)
Brief Title: Evaluation of the Safety and Effectiveness of the VRS100 System in PCI (ESSENCE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Raysight Intelligent Medical Technology Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other); West China Hospital (Other); Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VRS100 System
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases; Coronary Disease; Myocardial Ischemia; Arteriosclerosis; Vascular Disease Occlusive
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Coronary Disease; Myocardial Ischemia; Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRS100 robotic-assisted PCI (Experimental): VRS100 robotic-assisted PCI
  Interventions: Procedure: VRS100 robotic-assisted PCI
- Manual PCI (Active Comparator): Manual PCI
  Interventions: Procedure: Manual PCI

INTERVENTIONS:
Procedure: VRS100 robotic-assisted PCI — The VRS100 is intended for use in the remote delivery and manipulation of guidewires and rapid exchange balloon/stent catheters, and remote manipulation of guide catheters during percutaneous coronary intervention (PCI) procedures.
  Arms: VRS100 robotic-assisted PCI
Procedure: Manual PCI — Use the traditional technique of manually advancing intracoronary guidewires, balloons, and stents at the patient's tableside.
  Arms: Manual PCI

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the clinical and technical performance of the VRS100 system with disposable surgical kit in the delivery and manipulation of coronary guidewires and stent/balloon systems for use in percutaneous coronary interventions (PCI).

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria:

  1. Age ≥18 years.
  2. Patients with coronary artery disease undergoing Percutaneous Coronary Intervention (PCI).
  3. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
* Angiographic Inclusion Criteria:

  1. In situ primary coronary vascular disease.
  2. Reference vessel diameter is 2.5-4.0mm by visual estimate.
  3. Target lesion length is ≤30.0mm.
  4. Target lesion is a single de novo native coronary artery lesion. This lesion may consist of multiple lesions (with ≤10mm between diseased segments) and must be completely covered by a single stent with ≥5.0mm of normal segments on proximal and distal edges of the lesion.
  5. Target lesion diameter showing stenosis ≥70% by visual estimate, or ≥50% with myocardial ischemia.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded:

* General Exclusion Criteria:

  1. Subjects with indications for urgent PCI surgery.
  2. Evidence of an acute myocardial infarction within one week prior to the intended VRS100 procedure.
  3. Subject has undergone PCI within 72 hours prior to the VRS100 procedure.
  4. Subject has undergone PCI within 30 days prior to the VRS100 procedure and experienced a MACE or a serious adverse event (SAE).
  5. Severe heart failure (NYHA IV).
  6. Subject has suffered a stroke, or has an active peptic ulcer or upper gastrointestinal bleeding within 6 months prior to planned VRS100 procedure.
  7. Subject has known hypersensitivity or contraindication to aspirin, heparin, ticagrelor, clopidogrel, bivalirudin, PTX(paclitaxel), stainless steel, etc.
  8. Subject has acute or chronic kidney disease (serum creatinine level of >2.5 mg/dL or >221 umol/L) or need dialysis.
  9. Pregnant or breastfeeding, or planning to be pregnant.
  10. Repeated enrollment.
  11. Any other factors that the researchers consider not suitable for inclusion or completion of this study.
* Angiographic Exclusion Criteria:

  1. Any previous stent placement within 5.0 mm (proximal or distal) of the target lesion.
  2. The study lesion requires planned treatment with directional coronary atherectomy (DCA), laser, rotational atherectomy or any device except for balloon dilatation prior to stent placement.
  3. Cardiac allograft vasculopathy (CAV).
  4. The study vessel has evidence of intraluminal thrombus.
  5. Chronic total occlusion (CTO).
  6. The study lesion located in a native vessel distal to an ostial, bifurcation or anastomosis.
  7. Unprotected left main coronary artery disease defined as an obstruction greater than 50% diameter stenosis in the left main coronary artery.
  8. The study lesion or vessel proximal to the target lesion has severe tortuosity or calcification.
  9. Target lesion that cannot be fully covered by a single stent.
  10. more than 2 lesions requires treatment in one vessel.
  11. Subject requires treatment of more than one vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-09-08 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 48-hrs or hospital discharge, whichever occurs first
  Defined as angiographic success (residual stenosis after stenting of <30% with final TIMI [Thrombolysis In Myocardial Infarction] flow grade 3) without an in-hospital major adverse cardiovascular event (MACE) (cardiovascular death, MI, clinically driven target vessel revascularization).
Technical Success | 1 day
  Defined as the successful advancement and retraction of PCI devices using the VRS100 System and without conversion to manual operation.

SECONDARY OUTCOMES:
PCI Procedure Time | During procedure
  Defined as the time measured from the insertion of the guide catheter until the removal of the guide catheter.
Overall Procedure Time | During procedure
  Defined as the time measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
Fluoroscopy and/or X-Ray Time | During procedure
  As recorded by an X-Ray System utilized during the procedure.
Patient Radiation Exposure - Cumulative Dose | During procedure
  Cumulative dose (mGy) as recored during the procedure.
Contrast Fluid Volume | During procedure
  The amount of contrast fluid used (mL) during the procedure.
Performance of the Experimental Device | During procedure
  The frequency of failures and performance evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Study Director — Shanghai Zhongshan Hospital; Yong He, Principal Investigator — West China Hospital; Da Yin, Principal Investigator — Shenzhen People's Hospital
Locations (3):
- China (3):
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuang

IPD SHARING:
Plan to Share IPD: No